CLINICAL TRIAL: NCT01758107
Title: Study of Cyclosporine Withdrawal Regimen in Thai Renal Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Natavudh Townamchai, MD, MD, Chulalongkorn University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: monorapa
Record Dates: First submitted 2012-12-25; First posted 2013-01-01 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Renal Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus with Prednisolone (Experimental): Sirolimus with Prednisolone, and withdraw cyclosporine
  Interventions: Other: Withdraw cyclosporine
- Sirolimus with Cyclosporine with Prednisolone (No Intervention)

INTERVENTIONS:
Other: Withdraw cyclosporine
  Arms: Sirolimus with Prednisolone

SUMMARY:
Study safety of longterm immunosuppressive protocol with Sirolimus plus Prednisolone, and Calcineurin inhibitor withdrawal.

DETAILED DESCRIPTION:
Sirolimus with Cyclosporine minimization is the standard protocol for kidney transplantation in Chulalongkorn University. The investigators published the safety of this regimen in Transplantation Proceeding 2008; 40: 2206-8.

The investigators now further study in those patients who doing well with this regimen more than 1 year. The patients will be asked for kidney biopsy to evaluate and make sure they don't have subclinical rejection. The patients who don't have subclinical rejection will discontinue cyclosporine and continue with only sirolimus and prednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant with Sirolimus plus Cyclosporine plus Prednisolone more than 1 year

Exclusion Criteria:

* history of acute rejection, or subclinical rejection

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
longterm glomerular filtration rate defined by eGFR CKD-EPI | 5 years

SECONDARY OUTCOMES:
Acute rejection rate | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Bangkok, Thailand